CLINICAL TRIAL: NCT05289830
Title: A Phase II, Randomized, Double-blind, Trial Comparing Escitalopram to Placebo in Patients With Localized Pancreatic Cancer
Brief Title: Escitalopram to Placebo in Patients With Localized Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE6220
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Periampullary Cancer
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving Escitalopram (Experimental)
  Interventions: Drug: Escitalopram
- Participants receiving Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — Participants will receive Escitalopram 2 weeks: 10 mg/day (1 capsule) 8 weeks: 20 mg/day (2 capsules) 2 weeks: 10 mg/day (1 capsule)
  Arms: Participants receiving Escitalopram
Other: Placebo — Participants will receive placebo supplements 2 weeks: 1 capsule 8 weeks: 2 capsules 2 weeks: 1 capsule
  Arms: Participants receiving Placebo

SUMMARY:
Use of antidepressants for participants with localized pancreatic and periampullary cancer receiving neoadjuvant therapy.

DETAILED DESCRIPTION:
Anti-depressants have been shown to be beneficial in cancer participants. They reduce depressive symptoms and improve quality of life. Randomized trials have shown that antidepressants can reduce the development of depression in non-depressed participants with breast, melanoma, and head and neck cancers. It has been shown that treating depression can impact survival in cancer participants. Additionally, depressed pancreatic cancer participants have worse survival. Therefore, anti-depressants may also have implications for cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed localized or locally advanced pancreatic ductal adenocarcinoma or other periampullary adenocarcinoma (bile duct, duodenal, ampullary)
2. Subjects must not currently be on an antidepressant, anti-anxiety, anti-bipolar, or anti-psychotic medicine
3. Aged 18-80 years.
4. ECOG PS (Eastern Cooperative Oncology Group Performance Status) score of 0-2
5. Planned to have at least 12 weeks of neoadjuvant chemotherapy as standard of care cancer treatment
6. No diagnosis of bipolar disease
7. Willing to comply with all study procedures and be available for the duration of the study
8. Subjects must be mentally competent and must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients under the age of 18 or over 80
2. Metastatic pancreatic or other periampullary cancer
3. Resection of pancreatic cancer within the past year prior to study enrollment or planned surgery within the next 12 weeks.
4. Currently on an antidepressant, anti-anxiety, anti-bipolar or anti-psychotic medicine. Patients who have taken MAOIs (Monoamine Oxidase Inhibitors) within the past 6 months are excluded.
5. Patients with a history of seizure disorder
6. Patients with a recent medical history of myocardial infarction or unstable heart disease
7. Patients with a history of QTc prolongation or torsade de points, a baseline QTc

   1. interval of > 500ms, a history of drug-induced QTc prolongation or congenital long QT
   2. syndrome
8. Patients with Child-Pugh score of B or C
9. Patients with moderate to severe renal disease with a GFR (glomerular filtration rate) < 45.
10. Patients who cannot ingest oral medication
11. Patients with any history of mania
12. Known allergy to escitalopram
13. Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Winter, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
plan to publish the results
Supporting Information: CSR
Time Frame: 4 years to publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Receiving Escitalopram | Participants Receiving Placebo
Started | 2 | 2
Completed | 1 | 0
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Receiving Escitalopram | Participants Receiving Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the Rate of Depression
Description: Rate of depression will be measured using the Quick Inventory of Depressive Symptoms (QIDS) survey. This survey has 16 questions that are specific to the symptomatology of depression. Answers are given in the form of a four-point Likert scale ranging from 0-3, with zero relating to a standard sense of well-being and three correlating to the greatest feelings of depression. The survey is divided into 9 domains, and the survey is scored by adding the highest score on any one of the questions in each of the domains. Total scores range from 0 to 27, with greater scores indicating greater symptoms of depression.
Time Frame: 12 weeks from the start of treatment
Population: 1 participant in Arm 1 and 2 participants in Arm 2 were not evaluable at 12 weeks and did not complete the study
Measure: Number; unit: QIDS score
Arm/Group | Participants Receiving Escitalopram | Participants Receiving Placebo
Number analyzed (Participants) | 1 | 0
QIDS score | 13 |

2. Secondary Outcome: Quality of Life Using FACT-Hep (The Functional Assesment of Cancer Therapy-Hepatobiliary) Survey
Description: The FACT-Hep has 27 general questions and 18 questions that are specific to hepatopancreatobiliary cancer, for a total of 45 questions. The general questions span four domains: physical, social/family, emotional, and functional well-being 21. It requires less than 10 minutes to complete and targets the 6th-grade reading level. Answers are given in the form of a five-point Likert scale as follows: 0 (Not at all), 1 (A little bit), 2 (Somewhat), 3 (Quite a bit), and 4 (Very much). Points are re-calibrated and compiled, such that high scores indicate a higher quality of life. Scores range from 0 to 180.
Time Frame: Up to 12 weeks from the treatment date
Population: 1 participant in Arm 1 and 2 participants in Arm 2 were not evaluable at 12 weeks and did not complete the study
Measure: Number; unit: FACTS score
Arm/Group | Participants Receiving Escitalopram | Participants Receiving Placebo
Number analyzed (Participants) | 1 | 0
FACTS score | 90 |

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | Participants Receiving Escitalopram | Participants Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Escitalopram (N=2) | Participants Receiving Placebo (N=2)
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Escitalopram (N=2) | Participants Receiving Placebo (N=2)
Diarrhea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Creatinine increased (Investigations) | 1 | 0
Investigations, other- Creatinine clearance (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Slow accrual led to early termination. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT05289830/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT05289830/ICF_001.pdf